CLINICAL TRIAL: NCT04079946
Title: The Efficacy Of Complete Mesocolic Excision With Central Vessel Ligation Technique On Lymph Nodes And Safety Margins Compared With Conventional Surgery For Colon Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Essam Hassan Farghly, Resident Doctor At Assuit University Hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU93
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Cancer Colon
Keywords: cancer colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients for whom Complete mesocolic excision will be done (Active Comparator)
  Interventions: Procedure: Total Mesocolic Excision with Central Vessel Ligation
- patients had conventional surgery before (Active Comparator)
  Interventions: Procedure: conventional surgery of cancer colon

INTERVENTIONS:
Procedure: Total Mesocolic Excision with Central Vessel Ligation — sharp dissection of the anatomical layers and the dissection of the visceral plane from the parietal one . In addition a central division of the feeding arteries at their origins is performed at the level of superior mesenteric artery for tumors of the right colon and at the level of inferior mesenteric artery or the aorta for tumors of the left colon .this allows for removal of the maximum number of lymph nodes possible.
  Arms: patients for whom Complete mesocolic excision will be done
Procedure: conventional surgery of cancer colon — removal of the tumor with no ligation of the vessel centrally or removal of the whole mesocolon
  Arms: patients had conventional surgery before

SUMMARY:
Cancer Colon is one of the major public health problems worldwide. Complete eradication of the tumor with no recurrence or residual masses is a challenge which faces all the surgeons and medical staff all over the world. A lot of techniques were used to ensure 100 % eradication of the tumor and to cure the patients from cancer. Total Mesocolic Excision with Central Vessel Ligation is one of the recent techniques used for colon cancer surgeries. Here in the research the investigators answer the question of how this technique is superior and more beneficial in complete eradication of the tumor than the conventional surgery for colon cancer

ELIGIBILITY:
Inclusion Criteria:

* • Adult male and female Age of or above 18 years.

  * Tumor localization at the caecum, ascending colon, transverse colon, descending colon, sigmoid colon or rectosigmoid on preoperative endoscopy and radiographic imaging [barium enema or computed tomography (CT)]
  * No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease
  * Written informed consent

Exclusion Criteria:

* • Contraindications to major surgery and American Society of Anaesthesiologists (ASA) Physical Status scoring 4 which means extreme systemic disorders which have already become an eminent threat to life regardless of the type of treatment.

  * Infectious disease requiring treatment.
  * Pregnant women
  * Use of systemic steroids.
  * Severe pulmonary emphysema or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Lymph nodes harvest | Two years
  Number of retrieved lymph nodes can be extracted by this technique

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A. Hassanein, professor, Study Chair — Assiut University; Mohamed B. Kotb, profeesor, Study Director — Assiut University; Mahmoud T. Ahmed, lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol